CLINICAL TRIAL: NCT02967211
Title: A Twenty-six Week, Randomized, Open-label, 2-arm Parallel Group Real World Pragmatic Trial to Assess the Clinical and Health Outcomes Benefit of Transition to Toujeo Compared to "Standard of Care" Insulin in Basal Insulin Treated Patients With Uncontrolled Type 2 Diabetes Mellitus, With Six-Month Extension
Brief Title: A "Real World" Trial to Determine Efficacy and Health Outcomes of Toujeo Compared to "Standard of Care" Basal Insulin in Patients Already Using Basal Insulin
Acronym: REGAIN CONTROL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14060; 2015-001832-39 (EudraCT Number); U1111-1170-8132 (Other: UTN)
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin, Isophane; Isophane Insulin, Human; Insulin Detemir; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toujeo (Experimental): Toujeo will be administered once daily in addition to non-insulin antidiabetic agents
  Interventions: Drug: insulin glargine (U300)
- "Standard of care" commercially available basal insulin (Active Comparator): Lantus, Humulin Neutral Protamine Hagedorn (NPH), Levemir, and Tresiba or other basal insulin, including biosimilar insulin will be administered once or twice daily according to label in addition to non-insulin antidiabetic agents
  Interventions: Drug: insulin glargine (U100); Drug: NPH insulin; Drug: insulin detemir; Drug: insulin degludec

INTERVENTIONS:
Drug: insulin glargine (U300) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: HOE901; Toujeo
  Arms: Toujeo
Drug: insulin glargine (U100) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: HOE901; Lantus
  Arms: "Standard of care" commercially available basal insulin
Drug: NPH insulin — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Humulin NPH
  Arms: "Standard of care" commercially available basal insulin
Drug: insulin detemir — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Levemir
  Arms: "Standard of care" commercially available basal insulin
Drug: insulin degludec — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Tresiba
  Arms: "Standard of care" commercially available basal insulin

SUMMARY:
Primary Objective:

To demonstrate noninferiority of Toujeo versus "standard of care" basal insulin therapy as measured by glycated hemoglobin (HbA1c) change

Secondary Objectives:

* To demonstrate superiority of Toujeo versus "standard of care" basal insulin if non-inferiority criterion is met, measured by HbA1c change.
* To compare Toujeo to other "standard of care" basal insulin in terms of patient persistence with assigned basal insulin therapy with or without intensification.
* Risk of hypoglycemia including documented, symptomatic hypoglycemia (≤70 mg/dL) or severe (according to ADA Working Group).
* Change in fasting plasma glucose (FPG).
* Change in body weight.
* Differences in patient reported outcomes measured by Diabetes Treatment Satisfaction Questionnaire Status and Change versions (DTSQs and DTSQc).
* Change in hypoglycemic control subscale (HCS).
* Healthcare resource utilization including hospitalizations and emergency department or other health care provider visits and healthcare costs.

DETAILED DESCRIPTION:
The total study duration will be up to 55 weeks, consisting of a 1 week screening period at the site, a 26 week treatment period, and a 26 week extension period.

ELIGIBILITY:
Inclusion criteria :

* Patients with type 2 diabetes insufficiently controlled (HbA1c >7%) with current (≥6 months) "standard of care" basal insulin therapy (including insulin glargine U100, Levemir, NPH, or Tresiba) with or without oral agents (metformin, sulfonylurea, thiazolidinedione, DPP-4 inhibitor, SGLT-2 inhibitor, glinides, α glucosidase inhibitors) and with or without use of a GLP-1 receptor agonist.
* Fasting plasma glucose (FPG) >130 mg/dL (7.2 mmol/L).
* Adult patients who have signed Informed Consent Form (ICF) and privacy form(s).

Exclusion criteria:

* HbA1c ≤7%, no upper bound.
* Age <18 years.
* Type 1 diabetes mellitus.
* Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening, or any major systemic disease resulting in short life expectancy that in the opinion of the Investigator would restrict or limit the patient's successful participation for the duration of the study.
* Use of any product containing short or rapid acting insulin since the time of diagnosis with type 2 diabetes mellitus other than temporary use during a pregnancy or hospitalization.
* Use of any product containing short or rapid acting insulin occurring within 3 months prior to the time of screening.
* Use of oral hypoglycemic agents other than those noted in the inclusion criteria, GLP-1 receptor agonists not approved for use with insulin, or any investigational agent (drug, biologic, device) within 3 months prior to the time of screening.
* All contraindications to "standard of care" insulin therapy or warnings/precautions of use as displayed in the respective National Product labeling for these products.
* Hypersensitivity to insulin glargine or Toujeo excipients.
* Pregnancy or lactation.
* Women of childbearing potential with no effective contraceptive method.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2015-12-21; Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (percentage %) | Baseline to 6 months

SECONDARY OUTCOMES:
Proportion of patients who remain on assigned basal insulin therapy before intensification (persistent with assigned therapy) | At Month 6 and Month 12
Proportion of patients who remain on assigned basal insulin therapy whether intensification occurred or not | At Month 6 and Month 12
Proportion of patients who achieve target HbA1c (<6.5%, <7%, <7.5%, <8.0%) | At Month 6 and Month 12
Proportion of patients with HbA1c target (thresholds listed above) (attainment of metabolic benefit) without documented (blood glucose (BG) ≤70 mg/dl [3.9 mmol/L]) symptomatic or severe | At Month 6 and Month 12
Proportion of patients with HbA1c target (thresholds listed above) (attainment of metabolic benefit) without documented (BG <54 mg/dL, [3.0 mmol/L]) symptomatic or severe hypoglycemia | At Month 6 and Month 12
Change in HbA1c (percentage %) | Baseline, Month 12
Percentage of patients whose HbA1c decreased at least 0.5% | At Month 6 and Month 12
Percentage of patients whose HbA1c decreased at least 0.5% | At Month 6 and maintained at Month 12
Percentage of patients requiring intensification | At Month 6 and Month 12
Time to intensification | At Month 6 and Month 12
Change in fasting plasma glucose | From baseline to Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (118):
- Brazil (9):
  - Investigational Site Number 076-001, Curitiba
  - Investigational Site Number 076008, Fortaleza
  - Investigational Site Number 076004, Fortaleza
  - Investigational Site Number 076009, Rio de Janeiro
  - Investigational Site Number 076011, São José dos Campos
  - Investigational Site Number 076006, São Paulo
  - Investigational Site Number 076-003, São Paulo
  - Investigational Site Number 076005, São Paulo
  - Investigational Site Number 076010, Taguatinga
- Finland (6):
  - Investigational Site Number 246008, Helsinki
  - Investigational Site Number 246007, Muurame
  - Investigational Site Number 246002, Oulu
  - Investigational Site Number 246001, Oulu
  - Investigational Site Number 246009, Pori
  - Investigational Site Number 246004, Rauma
- France (14):
  - Investigational Site Number 250008, Amiens
  - Investigational Site Number 250011, Bordeaux
  - Investigational Site Number 250009, Caen
  - Investigational Site Number 250001, Corbeil-Essonnes
  - Investigational Site Number 250005, Eaubonne
  - Investigational Site Number 250026, La Rochelle
  - Investigational Site Number 250020, Montpellier
  - Investigational Site Number 250015, Mulhouse
  - Investigational Site Number 250003, Paris
  - Investigational Site Number 250010, Pierre-Bénite
  - Investigational Site Number 250014, Pierre-Bénite
  - Investigational Site Number 250025, Poitiers
  - Investigational Site Number 250002, Valenciennes
  - Investigational Site Number 250013, Vandœuvre-lès-Nancy
- Greece (4):
  - Investigational Site Number 300002, Athens
  - Investigational Site Number 300003, Kalamata
  - Investigational Site Number 300001, Lamia
  - Investigational Site Number 300004, Thessaloniki
- Ireland (2):
  - Investigational Site Number 372002, Dublin
  - Investigational Site Number 372003, Dublin
- Italy (23):
  - Investigational Site Number 380033, Arzignano (VI)
  - Investigational Site Number 380016, Catania
  - Investigational Site Number 380004, Catania
  - Investigational Site Number 380006, Catanzaro
  - Investigational Site Number 380031, Eboli
  - Investigational Site Number 380007, Forlì
  - Investigational Site Number 380018, Genova
  - Investigational Site Number 380020, Iglesias (CI)
  - Investigational Site Number 380015, Milan
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380012, Milan
  - Investigational Site Number 380011, Orbassano (TO)
  - Investigational Site Number 380026, Padua
  - Investigational Site Number 380021, Palermo
  - Investigational Site Number 380014, Partinico
  - Investigational Site Number 380032, Roma
  - Investigational Site Number 380002, Roma
  - Investigational Site Number 380023, Roma
  - Investigational Site Number 380036, San Benedetto del Tronto
  - Investigational Site Number 380024, Sarzana
  - Investigational Site Number 380013, Savigliano (CN)
  - Investigational Site Number 380017, Sesto S. Giovanni
  - Investigational Site Number 380025, Torino
- Romania (8):
  - Investigational Site Number 642008, Arad
  - Investigational Site Number 642005, Baia Mare
  - Investigational Site Number 642002, Brasov
  - Investigational Site Number 642006, Brasov
  - Investigational Site Number 642003, Cluj-Napoca
  - Investigational Site Number 642007, Cluj-Napoca
  - Investigational Site Number 642004, Târgu Mureş
  - Investigational Site Number 642001, Timișoara
- Spain (28):
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724019, Barcelona
  - Investigational Site Number 724012, Barcelona
  - Investigational Site Number 724011, Barcelona
  - Investigational Site Number 724027, Castellon
  - Investigational Site Number 724028, Córdoba
  - Investigational Site Number 724008, Galdakao (Bilbao)
  - Investigational Site Number 724010, León
  - Investigational Site Number 724001, Lleida
  - Investigational Site Number 724013, Madrid
  - Investigational Site Number 724018, Madrid
  - Investigational Site Number 724020, Málaga
  - Investigational Site Number 724025, Móstoles
  - Investigational Site Number 724006, Palma de Mallorca
  - Investigational Site Number 724007, Palma de Mallorca
  - Investigational Site Number 724024, Pontevedra
  - Investigational Site Number 724017, Sabadell
  - Investigational Site Number 724022, San Cristóbal de La Laguna - Santa Cruz de Tenerife
  - Investigational Site Number 724003, Sant Joan d'Alacant
  - Investigational Site Number 724030, Sant Joan Despí
  - Investigational Site Number 724023, Santa Cruz de Tenerife
  - Investigational Site Number 724014, Santiago de Compostela
  - Investigational Site Number 724005, Seville
  - Investigational Site Number 724016, Seville
  - Investigational Site Number 724004, Seville
  - Investigational Site Number 724021, Valencia
  - Investigational Site Number 724009, Valladolid
  - Investigational Site Number 724029, Vigo
- Switzerland (2):
  - Investigational Site Number 756003, Bern
  - Investigational Site Number 756002, Sankt Gallen
- United Kingdom (22):
  - Investigational Site Number 826033, Atherstone
  - Investigational Site Number 826016, Ayr
  - Investigational Site Number 826039, Blackburn
  - Investigational Site Number 826008, Bradford-on-Avon
  - Investigational Site Number 826004, Chertsey
  - Investigational Site Number 826038, Cornwall
  - Investigational Site Number 826031, Coventry
  - Investigational Site Number 826024, Darlington
  - Investigational Site Number 826035, Dudley
  - Investigational Site Number 826017, Glasgow
  - Investigational Site Number 826025, Huntingdon
  - Investigational Site Number 826002, Liverpool
  - Investigational Site Number 826018, Manchester
  - Investigational Site Number 826019, Manchester
  - Investigational Site Number 826037, Manchester
  - Investigational Site Number 826023, Norwich
  - Investigational Site Number 826009, Nuneaton
  - Investigational Site Number 826021, Plymouth
  - Investigational Site Number 826006, Portsmouth
  - Investigational Site Number 826020, Southampton
  - Investigational Site Number 826013, Taunton
  - Investigational Site Number 826007, Welwyn Garden City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- [Derived] Freemantle N, Mauricio D, Giaccari A, Bailey T, Roussel R, Franco D, Berthou B, Pilorget V, Westerbacka J, Bosnyak Z, Bonnemaire M, Cali AMG, Nguyen-Pascal ML, Penfornis A, Perez-Maraver M, Seufert J, Sullivan SD, Wilding J, Wysham C, Davies M. Real-world outcomes of treatment with insulin glargine 300 U/mL versus standard-of-care in people with uncontrolled type 2 diabetes mellitus. Curr Med Res Opin. 2020 Apr;36(4):571-581. doi: 10.1080/03007995.2019.1708287. Epub 2020 Jan 19. PMID 31865758